CLINICAL TRIAL: NCT06425224
Title: Effectiveness and Safety of Transcutaneous Posterior Tibial Nerve Stimulation Therapy for the Management of Patients With Premature Ejaculation. Phase III Clinical Trial
Brief Title: Effectiveness and Safety of TENS Therapy for Premature Ejaculation
Acronym: TENSPE2
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Boston Medical Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BMGC-M1
Record Dates: First submitted 2024-05-17; First posted 2024-05-22 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Premature Ejaculation; Sex Disorder; TEN
MeSH Terms: conditions — Premature Ejaculation; Sexual Dysfunction, Physiological | interventions — dapoxetine; Health Services Needs and Demand

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Group 1: Tens therapy + dapoxetine placebo on demand. (Active Comparator): There will be 3 weekly therapy sessions for 12 continuous weeks, lasting 30 minutes each. 20 Hertz with a pulse width of 200 µsec will be administered in each session. The intensity will be applied to each patient depending on individual tolerance. TENT therapy will be performed as follows:
  1. The active electrode is placed and adhered 3 - 5 cm above the internal malleolus and 1 cm behind the tibia.
  The second reference electrode is attached to the calcaneus.
  Continuous current, Frequency: 20 Hz Pulse width: 200 µsec, Time: 30 min. Intensity: to the patient's tolerance, gross motor perception to verify correct application, upon reaching it, increase the intensity to clearly sensory activation.
  They will also receive dapoxetine placebo (capsules with only excipients without active ingredient) as needed, taken 3 to 4 hours before sexual intercourse during the 12 weeks of the intervention.
  Interventions: Device: Tens therapy; Drug: Dapoxetine placebo
- Group 2: Standard treatment (dapoxetine 30 mg as needed) + placebo therapy. (Active Comparator): Patients in this group will receive dapoxetine 30 mg, taken 3 to 4 hours before sexual intercourse, for the 12 weeks of the study. In addition to the medication, patients will receive three weekly sessions of placebo therapy for twelve continuous weeks, lasting 30 minutes each. For this, the black electrode will be placed on the external malleolus and the red one 4 finger widths towards the head on the lateral edge of the tibia. 20 Hertz with a pulse width of 200 µsec will be administered in each session.
  Interventions: Drug: Standard treatment (dapoxetine 30 mg as needed); Device: Placebo therapy
- Group 3: Tens therapy + standard treatment (dapoxetine 30 mg as needed). (Experimental): Tens therapy + standard treatment (dapoxetine 30 mg as needed).
  Patients in this group will receive electrostimulation therapy of the posterior tibial nerve, 3 weekly therapy sessions for 12 continuous weeks, lasting 30 minutes each. 20 Hertz with a pulse width of 200 µsec will be administered in each session. The intensity will be applied to each patient depending on individual tolerance.
  In addition to the therapy, patients in this group will receive dapoxetine as needed, taken 3 to 4 hours before sexual intercourse during the 12 weeks of the intervention.
  Interventions: Device: Tens therapy; Drug: Standard treatment (dapoxetine 30 mg as needed)

INTERVENTIONS:
Device: Tens therapy — There will be 3 weekly therapy sessions for 12 continuous weeks, lasting 30 minutes each. 20 Hertz with a pulse width of 200 µsec will be administered in each session. The intensity will be applied to each patient depending on individual tolerance. TENT therapy will be performed as follows:
  1. The active electrode (cathode - red) is placed and adhered 3 - 5 cm above the internal malleolus and 1 cm behind the tibia.
  The second reference electrode (anode - black) is attached to the calcaneus.
  The equipment must previously be programmed under the following parameters:
  Continuous current Frequency: 20 Hz. Pulse width: 200 µsec Time: 30 min. Intensity: to the patient's tolerance, gross motor perception to verify correct application, upon reaching it, increase the intensity to clearly sensory activation.
  Arms: Group 1: Tens therapy + dapoxetine placebo on demand.; Group 3: Tens therapy + standard treatment (dapoxetine 30 mg as needed).
Drug: Dapoxetine placebo — Patients in this group will receive dapoxetine placebo (capsules with only excipients without active ingredient) as needed, taken 3 to 4 hours before sexual intercourse during the 12 weeks of the intervention.
  Arms: Group 1: Tens therapy + dapoxetine placebo on demand.
Drug: Standard treatment (dapoxetine 30 mg as needed) — Patients in this group will receive dapoxetine 30 mg, taken 3 to 4 hours before sexual intercourse, for the 12 weeks of the study
  Arms: Group 2: Standard treatment (dapoxetine 30 mg as needed) + placebo therapy.; Group 3: Tens therapy + standard treatment (dapoxetine 30 mg as needed).
Device: Placebo therapy — In addition to the medication, patients will receive three weekly sessions of placebo therapy for twelve continuous weeks, lasting 30 minutes each. For this, the black electrode will be placed on the external malleolus and the red one 4 finger widths towards the head on the lateral edge of the tibia. 20 Hertz with a pulse width of 200 µsec will be administered in each session.
  Arms: Group 2: Standard treatment (dapoxetine 30 mg as needed) + placebo therapy.

SUMMARY:
The objective of this clinical trial is to evaluate the effectiveness and safety of transcutaneous posterior tibial nerve stimulation therapy in patients with premature ejaculation. The main question to answer is:

Can the effectiveness and safety of transcutaneous electrostimulation of the posterior tibial nerve alone and combined with standard pharmacological treatment be evaluated in men with lifelong premature ejaculation, compared to standard pharmacological treatment with dapoxetine?

Patients will:

Be randomized in acontrolled clinical trial. Patients with a diagnosis of premature ejaculation who attend Boston Medical Group clinics in Mexico City will be included.

Be assigned by randomization to one of three treatment groups:

* Group 1: Tens therapy + dapoxetine placebo on demand.
* Group 2: Standard treatment (dapoxetine 30 mg as needed) + placebo therapy.
* Group 3: Tens therapy + standard treatment (dapoxetine 30 mg as needed).

ELIGIBILITY:
Inclusion Criteria:

* Primary premature ejaculation according to the definition of the International Society for Sexual Medicine (ISSM-International Society for Sexual Medicine) (30): a) ejaculation always or almost always occurs within the first minute after penetration, b) inability to delay ejaculation in all or almost all penetrations, c) negative personal consequences are generated, such as stress, annoyance, frustration and/or avoidance of sexual intimacy.
* Age between 18 and 62 years.
* PEDT score greater than 11.
* Stable heterosexual relationship for at least 6 months with interest in maintaining it for at least the duration of the study.
* Sexual activity at least once a week.
* Minimum chronicity of PD of 6 months.
* Voluntary participation in the study.
* Signing of the informed consent prior to participation in the study.

Exclusion Criteria:

* IIEF-EF score less than 26.
* Glaucoma
* Clinically significant comorbidity: cardiovascular, hepatic, thromboembolic, neurological, locomotor, endocrine, oncological, renal or rheumatological.
* History of retroperitoneal surgery, radiotherapy or multiple sclerosis.
* History of mental illness: depression, anxiety, suicidal behavior, bipolar disorder, agoraphobia, dysthymia, social phobia, obsessive-compulsive disorder, post-traumatic stress disorder, psychiatric disorder, reported by the patient or due to the use of a medication for one of these conditions.
* Consumption of medications that affect ejaculatory control such as psychiatric medications, opioid analgesics, alpha blockers.
* Treatment for PE in the last 3 months.
* Treatment for epileptic syndromes or Parkinson's disease.
* Use of pacemaker or cardiac defibrillator.
* Skin lesions in the area where the electrodes are placed.
* Abuse or dependence on psychoactive substances: alcohol, hallucinogenic drugs.
* Couple who are pregnant or interested in conceiving a pregnancy in the next 3 months.

Ages: 18 Years to 62 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 129 (Estimated)
Dates: Start 2022-06-15 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Change in intravaginal latency time | 12 weeks
  Average change in intravaginal latency time, measured with a stopwatch by the couple.

SECONDARY OUTCOMES:
Change in intravaginal latency time | 24 weeks
  Average change in intravaginal latency time, measured with a stopwatch by the couple.
Clinical improvement in premature ejaculation | At weeks 12 (end of therapy) and 24 (three months of follow-up).
  Proportion of patients with clinical improvement in premature ejaculation, defined as a three-fold increase in the intravaginal ejaculatory latency time.
Change in the diagnosis of premature ejaculation | At weeks 12 and 24 (greater than 12 to less than 12).
  Proportion of patients with a change in the diagnosis of premature ejaculation according to the PEDT (Premature Ejaculation Diagnostic Tool) questionnaire score in the intervention groups
Global Impression of Change Scale | Weeks 12 and 24.
  Global Impression of Change Scale score
PEP (Premature Ejaculation Profile) questionnaire score | At weeks 12 and 24
  Change in the PEP (Premature Ejaculation Profile) questionnaire score
Adverse events | 24 weeks
  Type, frequency and severity of adverse events during therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Barba, MD, Principal Investigator — Boston Medical Group
Locations (1):
- Boston Medical Group, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No